CLINICAL TRIAL: NCT00752531
Title: Evaluation of Home Automated Telemanagement in COPD
Brief Title: Effectiveness of Home Automated Telemanagement in Chronic Obstructive Pulmonary Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 596; R01HL071690 (NIH); R01HL071690-01 (NIH)
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HAT (Experimental)
  Interventions: Behavioral: Home Automated Telemanagement (HAT)
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Home Automated Telemanagement (HAT) — The HAT was designed as an Internet-based telemedicine system that (1) provides ongoing education to patients about their chronic disease, (2) helps patients follow their self-care plans, and (3) helps health care practitioners monitor their patients' self-management processes according to current clinical guidelines. During each telecommunication session, patients perform self-testing and receive structured disease-specific education, patient-tailored counseling, and advice on how to follow their individual self-care plans based on the current results of self-testing.
  Other Names: HAT
  Arms: HAT

SUMMARY:
All chronic obstructive pulmonary diseases (COPDs) block air flow to the lungs, and the two most common forms, emphysema and chronic bronchitis, are the most common causes of respiratory failure. Previous research shows that if COPD patients know more about their disease and how to manage it themselves, they will improve their quality of life and reduce their need for urgent care. However, traditional methods of teaching COPD patients about their disease and self-management skills are expensive and require intensive work. A new, less expensive way of reaching a large group of people with this information is needed to help patients stay healthier and happier with their treatment. This study will create a computer program that can help people learn about their disease and how to manage it themselves. This study will then determine whether the computer program, called Home Automated Telemanagement (HAT), helps patients with COPD in managing their disease and following their treatment plans.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is the result of damage to the lungs, making it hard for someone with COPD to breathe. The two most common forms of COPD are emphysema and chronic bronchitis, which can cause respiratory failure and irreversible damage to the lungs. There is no cure for COPD, but interventions that help patients understand their disease and how to manage it themselves can improve patient quality of life and prevent crises that would require urgent care. The National Heart, Lung, and Blood Institute and World Health Organization's Global Health Initiative for Chronic Obstructive Lung Disease (GOLD) recommend multiple components for maintaining care of patients with COPD, including regular patient assessment, education concerning COPD, effective communication between patients and their health care providers, patient compliance with treatment plans, implementation of behavioral change models for increasing health, and social support for patients and caregivers. Evidence suggests that these guidelines are not used widely, possibly because they are labor intensive and expensive and require frequent visits to a medical facility. Because effective interventions are not being used by patients and because previous studies show telecommunication technologies are successful in patient self-care, this study will develop a home automated telemanagement (HAT) system incorporating many of the GOLD guidelines for use in patients' homes.

HAT will be an Internet-based system providing ongoing education for patients about COPD, helping patients follow their self-care plans, and helping health care providers monitor patients' self-management through daily access. The system will consist of three pieces: (1) patient units that include a computer or palmtop Internet accessible device equipped with a disease-specific testing device, (2) a HAT server to analyze and store self-testing results, and (3) clinician units that can review patient results on the Internet. By incorporating text, audio, and visual components, the system will provide advice on self-care plans tailored to each patient and will notify health care providers of each patient's plan compliance.

This study has two phases. In the first, a HAT system for COPD will be refined based on user interviews and focus groups. In the second, researchers will test its effectiveness in keeping people with COPD healthy and ensuring they follow their self-care plans.

During the second phase of the study, which will last 18 months, all participants will be provided with an Internet-capable computer. All participants will continue seeing their own doctors and following a regular treatment plan prescribed by their doctors. Some will be randomly assigned to also receive the HAT system. Those given the HAT system will take a 1-hour training course on its use and be expected to use it daily for a 10- to 15-minute self-assessment and disease diary entry. The HAT system will also have other assessment, counseling, and education tools that participants can use. Participants will be assessed seven times, with four assessments at the research site and three at the home of each participant. Assessments will be conducted every 3 months, with those at the research site scheduled at baseline and Months 6, 12, and 18. Participants will complete questionnaires and be interviewed at each assessment to measure the severity of their disease, well-being, and attitudes toward the disease. During the assessments at the research site, additional tests in breathing and physical fitness will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of chronic obstructive pulmonary disorder (COPD)
* Moderate to severe COPD according to NHLBI/WHO Global Initiative for Chronic Obstructive Lung Disease (GOLD) classification (Stages II to III)
* Understands spoken English
* Has a functional telephone line or cable at home

Exclusion Criteria:

* Evidence that the participant may move from the study area before the completion of the study
* Presence of any health condition that would preclude participation, such as a psychiatric diagnosis or physical disability that would severely affect a participant's ability to carry out study procedures
* Inability to use telephone unassisted

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2003-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Clinical health, including lung function and respiratory symptoms | Measured at baseline and every 3 months for 18 months

SECONDARY OUTCOMES:
Disease-specific quality of life | Measured at baseline and every 3 months for 18 months
Exercise tolerance | Measured at baseline and at Months 6, 12, and 18
Urgent health care utilization | Measured at baseline and every 3 months for 18 months
Self-efficacy for COPD patients | Measured at baseline and every 3 months for 18 months
Activities of daily living (ADL) | Measured at baseline and every 3 months for 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Finkelstein, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633